CLINICAL TRIAL: NCT07061886
Title: Drug Effects on Mood and Behavior - Expectancy
Acronym: MESA-X
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB25-0658; 5R01DA002812-35 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: LSD
Keywords: Healthy Adults
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LSD (13 micrograms), Identity of substance known (Experimental): LSD tartrate in tasteless solution (0.13 mL). Subjects will receive LSD, and they (but not the research assistant) will be told the identity of the drug.
  Interventions: Drug: LSD
- LSD (13 micrograms), Identity uncertain (Active Comparator): LSD tartrate in tasteless solution (0.13 mL). Subjects will be told they might receive a stimulant, sedative, low dose of hallucinogen, or placebo, and will receive LSD.
  Interventions: Drug: LSD
- Placebo, Identity of substance known (Placebo Comparator): Distilled water (0.13 mL). Subjects will receive placebo, and they (but not the research assistant) will be told the identity of the drug.
  Interventions: Drug: Placebo
- Placebo, Identity uncertain (Placebo Comparator): Distilled water (0.13 mL). Subjects will be told they might receive a stimulant, sedative, low dose of hallucinogen, or placebo, and will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LSD — The serotonin 2A receptor agonist LSD
  Other Names: Lysergic acid diethylamide
  Arms: LSD (13 micrograms), Identity of substance known; LSD (13 micrograms), Identity uncertain
Drug: Placebo — Distilled water (0.26 mL)
  Arms: Placebo, Identity of substance known; Placebo, Identity uncertain

SUMMARY:
This study will examine the effects of a single low dose of the 5HT2A agonist LSD (Lysergic Acid Diethylamide) (13 µg) or placebo in individuals who are or are not explicitly told what drug they will receive. Although it is known that expectancies strongly influence subjective responses to most drugs, no studies have examined expectancies on response to a very low dose of LSD. This is especially important in the context of 'microdosing' of drugs. People who practice microdosing typically do so with strong expectations of positive effects, making it difficult to determine whether there is a pharmacological effect. To minimize expectancies in the laboratory, participants are usually not told exactly what drug they will receive (i.e., double-blind), but given a range of possibilities. In the present study, the study team will test half the subjects under single-blind conditions, where the participants (but not the research assistant) will know exactly what they are receiving. Other subjects will receive the usual instructions. Healthy volunteers will receive either a marginally detectable dose of LSD (13 micrograms) or placebo, under conditions where they i) know for sure what drug they are receiving or ii) where the identity of the drug is uncertain. Four groups of subjects (N=12 each) will attend single 4-hour laboratory session. The study team will examine subjective and behavioral responses to the drug in each of four conditions (Known-Drug; Known-Placebo; Uncertain-Drug; Uncertain-Placebo).

DETAILED DESCRIPTION:
Expectancies are known to influence responses to psychoactive drugs. The study team and others have shown previously, using a balanced placebo design, that expectancies influence responses to alcohol, nicotine, caffeine, stimulant drugs, and cannabinoids. In these studies subjects are randomly assigned to one of four conditions: Expect the drug and get the drug; Expect the drug and get placebo; Expect placebo and get the drug; Expect placebo and get placebo. This allows researchers to separate pharmacological effects from expectancy effects.

Recently there has been much discussion about the role of expectancies specifically in responses to psychedelic drugs. Expectancies are especially important in the use of very low doses, referred to as 'microdoses'. These doses are typically at or below the threshold of detectability, but users take them with strong prior beliefs that the drugs improve mood and cognition. The beneficial effects have been difficult to demonstrate under laboratory conditions, perhaps because in the laboratory the drugs are administered without the explicit expectation of benefits, and the administration of the drugs is to some extent blinded. The present study is designed to separate the pharmacological effects of a low dose of LSD from effects that are influenced by expectancies.

ELIGIBILITY:
Inclusion Criteria:

* English Fluency
* High school education or higher
* BMI between 19-30 kg/m2

Exclusion Criteria:

* Individuals with a medical condition contraindicating study participation as determined by the study physician (e.g., liver disease, abnormal EKG, liver or cardiovascular disease)
* High blood pressure (>140/90)
* Current suicidal ideation or suicide attempt in past 12 months
* Past year severe substance use disorder
* Personal or first-degree relative with history of psychosis
* Currently taking any psychiatric medication (for conventional antidepressants must be off for ≥ 2 weeks)
* Active panic disorder
* Severe obsessive-compulsive disorder
* Severe post-traumatic stress disorder
* Women who are pregnant or planning to become pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | During in-lab session: Pre-drug, and every 60 minutes post-drug from 0-4 hours
  Momentary states will be assessed using VAS to measure ratings of 'depressed', 'anxious', 'motivated', and 'energetic', on a scale of 0 (Not at all) to 100 (Very much).
Addiction Research Center Inventory (ARCI) | During in-lab session: Pre-drug, and every 60 minutes post-drug from 0-4 hours
  The ARCI is a 53-item true or false questionnaire that assess effects of specific drug classes. It includes scales measuring: amphetamine (A); benzedrine group (BG; energy and intellectual efficiency); morphine-benzedrine group (MBG; euphoric effects); LSD (hallucinogen-like effects); pentobarbital-chlorpromazine-alcohol group (PCAG; sedative effects); and marijuana (M).
Drug Effects Questionnaire (DEQ) | During in-lab session: Pre-drug, and every 60 minutes post-drug from 0-4 hours
  The DEQ measures overall drug effects. It consists of questions on a visual analog scale about the subjective effects of drugs. Subjects are asked to rate the extent they feel a drug effect, whether they like or dislike the drug effect, and if given a choice would they want to take more of the drug. Scores range from 0-100.
5 Dimensions of Altered States of Consciousness (5D-ASC) scale | End of session (4 hours post-drug)
  The 5D-ASC assesses altered states of consciousness in five domains, and is sensitive to LSD administration (Schmid et al. 2014). Scores range from 0-100.
Ultimatum Game | During in lab session: 1.5 hours post-drug
  In this task, participants play the role of responder in a series of single-shot computer interactions. They engage in 60 trials in which they interact with different computer-simulated proposers. On each trial they are allocated $10 to split between themselves and the participant. Participants will receive 60 different monetary offers ranging from fair (50:50 splits) to increasingly unfair (10:90 splits), presented in random order. For each offer, participants must decide whether to accept the offer, in which case both players receive the proposed amounts, or reject the offer, in which case both players receive nothing. This task will measure how the drug affects perception of fairness, and decision-making in social contexts. The task takes approximately a 30 minutes to complete.

SECONDARY OUTCOMES:
Cardiovascular (Heart rate, blood pressure) | During in-lab session: baseline (pre-drug), and every 60 minutes post-drug from 0-4 hours
  Systolic pressure (SP), diastolic pressure (DP) and heart rate (HR) will be measured using a portable digital blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Molla, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aron, A., Melinat, E., Aron, E. N., Vallone, R. D., & Bator, R. J. (1997). The Experimental Generation of Interpersonal Closeness: A Procedure and Some Preliminary Findings. Personality and Social Psychology Bulletin, 23(4), 363-377. https://doi.org/10.1177/0146167297234003
- [Background] Beck, A. T., Steer, R. A., & Brown, G. (1996). Beck Depression Inventory-II (BDI-II). In APA PsycTests
- [Background] Bershad AK, Schepers ST, Bremmer MP, Lee R, de Wit H. Acute Subjective and Behavioral Effects of Microdoses of Lysergic Acid Diethylamide in Healthy Human Volunteers. Biol Psychiatry. 2019 Nov 15;86(10):792-800. doi: 10.1016/j.biopsych.2019.05.019. Epub 2019 Jun 3. PMID 31331617
- [Background] de Wit H, Molla HM, Bershad A, Bremmer M, Lee R. Repeated low doses of LSD in healthy adults: A placebo-controlled, dose-response study. Addict Biol. 2022 Mar;27(2):e13143. doi: 10.1111/adb.13143. Epub 2022 Feb 1. PMID 35106880
- [Background] Dittrich A. The standardized psychometric assessment of altered states of consciousness (ASCs) in humans. Pharmacopsychiatry. 1998 Jul;31 Suppl 2:80-4. doi: 10.1055/s-2007-979351. PMID 9754838
- [Background] Fadiman, J and Gruber, J (2025) Microdosing for Health, Healing, and Enhanced Performance, St Martins Group
- [Background] Fischman MW, Foltin RW. Utility of subjective-effects measurements in assessing abuse liability of drugs in humans. Br J Addict. 1991 Dec;86(12):1563-70. doi: 10.1111/j.1360-0443.1991.tb01749.x. PMID 1786488
- [Background] Güth, W, RSchmittberger, B Schwarze (1982) An experimental analysis of ultimatum bargaining. Journal of Economic Behavior & Organization, Volume 3, 367-388
- [Background] Hammami MM, Al-Gaai EA, Alvi S, Hammami MB. Interaction between drug and placebo effects: a cross-over balanced placebo design trial. Trials. 2010 Nov 19;11:110. doi: 10.1186/1745-6215-11-110. PMID 21092089
- [Background] Lyvers MF, Maltzman I. The balanced placebo design: effects of alcohol and beverage instructions cannot be independently assessed. Int J Addict. 1991 Sep;26(9):963-72. doi: 10.3109/10826089109058933. PMID 1743824
- [Background] Martin WR, Sloan JW, Sapira JD, Jasinski DR. Physiologic, subjective, and behavioral effects of amphetamine, methamphetamine, ephedrine, phenmetrazine, and methylphenidate in man. Clin Pharmacol Ther. 1971 Mar-Apr;12(2):245-58. doi: 10.1002/cpt1971122part1245. No abstract available. PMID 5554941
- [Background] McNair, D., Lorr, M., Droppleman, L., (1971). POMS, Profile of Mood States. E. a. I. T. Services.
- [Background] Metrik J, Kahler CW, Reynolds B, McGeary JE, Monti PM, Haney M, de Wit H, Rohsenow DJ. Balanced placebo design with marijuana: pharmacological and expectancy effects on impulsivity and risk taking. Psychopharmacology (Berl). 2012 Oct;223(4):489-99. doi: 10.1007/s00213-012-2740-y. Epub 2012 May 16. PMID 22588253
- [Background] Molla H, Lee R, Tare I, de Wit H. Greater subjective effects of a low dose of LSD in participants with depressed mood. Neuropsychopharmacology. 2024 Apr;49(5):774-781. doi: 10.1038/s41386-023-01772-4. Epub 2023 Dec 2. PMID 38042914
- [Background] Murphy RJ, Muthukumaraswamy S, de Wit H. Microdosing Psychedelics: Current Evidence From Controlled Studies. Biol Psychiatry Cogn Neurosci Neuroimaging. 2024 May;9(5):500-511. doi: 10.1016/j.bpsc.2024.01.002. Epub 2024 Jan 26. PMID 38280630
- [Background] Palmer AM, Brandon TH. Nicotine or expectancies? Using the balanced-placebo design to test immediate outcomes of vaping. Addict Behav. 2019 Oct;97:90-96. doi: 10.1016/j.addbeh.2019.04.026. Epub 2019 Apr 26. PMID 31174168
- [Background] Skopp G, Potsch L, Mattern R, Aderjan R. Short-term stability of lysergic acid diethylamide (LSD), N-desmethyl-LSD, and 2-oxo-3-hydroxy-LSD in urine, assessed by liquid chromatography-tandem mass spectrometry. Clin Chem. 2002 Sep;48(9):1615-8. No abstract available. PMID 12194952
- [Background] Szigeti B, Heifets BD. Expectancy Effects in Psychedelic Trials. Biol Psychiatry Cogn Neurosci Neuroimaging. 2024 May;9(5):512-521. doi: 10.1016/j.bpsc.2024.02.004. Epub 2024 Feb 20. PMID 38387698
- See also: Bershad et al., 2019 — http://doi.org/10.1016/j.biopsych.2019.05.019
- See also: Dittrich, 1998 — http://doi.org/10.1055/s-2007-979351
- See also: Hammami et al., 2010 — http://doi.org/10.1186/1745-6215-11-110
- See also: Metrik et al., 2012 — http://doi.org/10.1007/s00213-012-2740-y
- See also: Molla et al., 2024 — http://doi.org/10.1038/s41386-023-01772-4
- See also: Murphy et al., 2024 — http://doi.org/10.1016/j.bpsc.2024.01.002
- See also: Palmer et al., 2019 — http://doi.org/10.1016/j.addbeh.2019.04.026
- See also: Szigeti & Heifets, 2024 — http://doi.org/10.1016/j.bpsc.2024.02.004